CLINICAL TRIAL: NCT02640417
Title: Avaliação clínica-terapêutica Comparativa em Lombalgias de Etiologia Traumato-compressivas Utilizando-se Vitaminas do Complexo B e nucleotídeos
Brief Title: Nucleotides and B Vitamins in the Treatment of Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Responsible Party: Principal Investigator, Marco Antonio Naslausky Mibielli, Professor and Chairman of Orthopedics, Fundação Educacional Serra dos Órgãos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NHCN-03-12-15
Record Dates: First submitted 2015-12-15; First posted 2015-12-29 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Low Back Pain
Keywords: Nucleotides (uridine, cytidine); Vitamin B1; Vitamin B6; Vitamin B12
MeSH Terms: conditions — Low Back Pain | interventions — Nucleotides; Vitamin B 12; Vitamin B Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nucleotides + B12 (Experimental): Nucleotides + Vitamin B12 Dose: two capsules, three times per day + placebo corresponding to Group B treatment
  Interventions: Drug: Nucleotides + B12
- B vitamins (Active Comparator): Vitamin B1 + Vitamin B6 + Vitamin B12 Dose: one tablet, three times daily + placebo corresponding to Group A treatment
  Interventions: Drug: B Vitamins

INTERVENTIONS:
Drug: Nucleotides + B12 — Oral treatment with either Nucleotides + Vitamin B12
  Other Names: Group A
  Arms: Nucleotides + B12
Drug: B Vitamins — Oral treatment with vitamins B1, B6, and B12
  Other Names: Group B
  Arms: B vitamins

SUMMARY:
This is a double-blind, randomized study in parallel groups of subjects presenting with low back pain. Randomized subjects will receive treatment for 60 days with either a combination of nucleotides and vitamin B12 or vitamin B1+B6+B12.

DETAILED DESCRIPTION:
This is a double-blind, randomized study in parallel groups of subjects presenting with low back pain. Randomized subjects will receive treatment for 60 days with either a combination of nucleotides and vitamin B12 or vitamin B1+B6+B12. The aim of this study is to evaluate and compare the therapeutic effect of the combination of nucleotides + vitamin B12 with that of the combination of vitamins B1, B6 and B12 in low back pain. Safety and efficacy will be monitored throughout the treatment period. Subjects will be randomized in a double-blind fashion to either treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, at least 18 years of age
* Clinical presentation of acute lumbago (<3 days of initial visit, with and without functional alteration, with medium intensity: Visual Analog Pain score between 20mm and 80mm
* Female subjects should be post-menopausal or using birth control
* Subjects must sign informed consent document

Exclusion Criteria:

* Intolerance to any component of the study treatments
* Pregnancy or breastfeeding
* Need for surgical treatment
* Use of other analgesic drugs
* dyshematopoiesis or coagulation disorder
* Gastric or intestinal ulcer
* Gastrointestinal, cerebrovascular, or other bleeding
* Creatinine >3x% reference range
* Urea, ALT, AST, or GGT >2x% reference range
* Any other disease or condition that in the investigator's opinion should exclude the subject from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Adverse Event Occurrence | Throughout 60 day treatment period
  Percentage of subjects in each treatment group presenting with adverse events

SECONDARY OUTCOMES:
Low back pain Questionnaire | Pretreatment, Visit 2 (at 30 days of treatment), Visit 3 (at 60 days of treatment)
  Percentage of subjects in each treatment group presenting improvement of >5 points in Questionnaire scores
Visual Analog Pain Scores | Pretreatment, Visit 2 (at 30 days of treatment), Visit 3 (at 60 days of treatment)
  Percentage of subjects in each treatment group presenting improvement of VAS pain scores in relation to pretreatment
Finger-to-Floor Distance | Pretreatment, Visit 2 (at 30 days of treatment), Visit 3 (at 60 days of treatment)
  Percentage of subjects in each treatment group presenting improvement of >3cm in finger to floor distance in relation to pretreatment values

CONTACTS AND LOCATIONS:
Overall Officials: Marco AN Mibielli, MD, Principal Investigator — UNIFESO - Fundação Educacional Serra dos Órgãos